CLINICAL TRIAL: NCT00391417
Title: Phase III, Multicenter, Double-Blind Study of the Safety and Efficacy of Bio-E-Gel (Topical Estradiol Gel) Versus Placebo for Treatment of Vasomotor Symptoms and Vulvovaginal Atrophy in Postmenopausal Females
Brief Title: Efficacy and Safety of a Topical Estradiol Gel for Treatment of Postmenopausal Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioSante Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EST005
Record Dates: First submitted 2006-10-20; First posted 2006-10-24 (Estimated); Last update posted 2006-10-24 (Estimated); Status verified 2006-10

CONDITIONS: Hot Flashes
Keywords: hot flush; hot flash; estrogen; vaginal atrophy
MeSH Terms: conditions — Hot Flashes

INTERVENTIONS:
Drug: estradiol gel

SUMMARY:
The purpose of this study is to determine the efficacy and safety of a topical estradiol gel for the treatment of hot flushes in postmenopausal women.

DETAILED DESCRIPTION:
Estrogens are a group of hormones that play an important role in normal sexual and reproductive development in women. Estrogens serve many functions in the body. They stimulate oocyte maturation and endometrial growth, decrease bone resorption, initiate the development of secondary sex characteristics, maintain reproductive organs and glands, and affect the activity of the central nervous system. At menopause, the decrease in estrogen concentrations is often accompanied by vascular instability (hot flushes and night sweats), a rise in the incidence of heart disease, and an increasing rate of bone loss. Estrogen is available as an oral drug, a transdermal patch, or as a gel or lotion. Transdermal estrogen is preferable as compared to oral, since it avoids the first-pass metabolism in the liver. Since release of the WHI findings, current treatment recommendations are for the lowest effective dose for the shortest period of time to treat postmenopausal symptoms.

Comparison: Three doses of a transdermal estradiol gel as compared to placebo for the treatment of vasomotor and vulvovaginal atrophy symptoms in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* serum estradiol level less than or equal to 20 pg per mL
* serum FSH greater than 40 mIU per mL

Exclusion Criteria:

* Pathological cancer findings on screening
* abnormal endometrium
* serious hepatic, renal or cardiac disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 431
Dates: Start 2003-09; Study Completion 2005-04

PRIMARY OUTCOMES:
Mean change from baseline in number of daily moderate to severe hot flushes.
Mean change from baseline in daily hot flush severity.
Mean change from baseline in vulvovaginal atrophy symptoms.

SECONDARY OUTCOMES:
Percent change from baseline in daily moderate to severe hot flush rates over time.
Percent change from baseline in hot flush severity over time.
Proportion of subjects with fifty to one hundred percent reductions in daily moderate to severe hot flushes.
Proportion of subjects with fifty to one hundred percent reductions in hot flush severity
Mean change from baseline in subject vaginal health self assessment over time.
Mean change from baseline in physician assessment of vaginal atrophy.

REFERENCES:
- [Derived] Simon JA, Bouchard C, Waldbaum A, Utian W, Zborowski J, Snabes MC. Low dose of transdermal estradiol gel for treatment of symptomatic postmenopausal women: a randomized controlled trial. Obstet Gynecol. 2007 Mar;109(3):588-96. doi: 10.1097/01.AOG.0000254160.62588.41. PMID 17329509